CLINICAL TRIAL: NCT03713255
Title: Analgesic Benefits of the Novel Mid-point Transverse Process to Pleura (MTP) Block for Ambulatory Breast Cancer Surgery: A Randomized Controlled Trial
Brief Title: Mid-point Transverse Process to Pleura Block for Breast Cancer Surgery: A Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20180259-01H
Record Dates: First submitted 2018-09-27; First posted 2018-10-19 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Breast Cancer; Acute Pain; Anesthesia
Keywords: Regional Anesthesia; Paravertebral Block; Breast Cancer Surgery; MTP block
MeSH Terms: conditions — Breast Neoplasms; Acute Pain | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, quadruple-blinded, three arm parallel group clinical trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (participant, care provider, investigator, outcomes assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PVB group (Active Comparator): paravertebral blocks with 0.5% ropivacaine and epinephrine 2.5 mcg/mL
  Interventions: Procedure: PVB group
- MTP block group (Experimental): MTP blocks with 0.5% ropivacaine and epinephrine 2.5 mcg/mL
  Interventions: Procedure: MTP block group
- control group (Sham Comparator): local anesthetic infiltration subcutaneous 1% lidocaine
  Interventions: Procedure: Control Group

INTERVENTIONS:
Procedure: PVB group — Patients in this group will receive preoperative ultrasound-guided thoracic paravertebral block using ropivacaine 0.5% with epinephrine 2.5 mcg/mL, and supplemental standardized anesthetic/analgesic regimen (Acetaminophen / NSAIDs / opioids for breakthrough pain).
  Arms: PVB group
Procedure: MTP block group — Patients in this group will receive preoperative ultrasound-guided mid-point transverse process to pleura block using ropivacaine 0.5% with epinephrine 2.5 mcg/mL, and supplemental standardized anesthetic/analgesic regimen (Acetaminophen / NSAIDs / opioids for breakthrough pain).
  Arms: MTP block group
Procedure: Control Group — Patients in this group will receive preoperative ultrasound-guided sham block with subcutaneous local anesthetic injection using lidocaine 1%, and supplemental standardized anesthetic/analgesic regimen (Acetaminophen / NSAIDs / opioids for breakthrough pain).
  Arms: control group

SUMMARY:
This study will compare the analgesic effects of midpoint transverse process to pleura (MTP) block to control as well as thoracic paravertebral block.

DETAILED DESCRIPTION:
Paravertebral blocks (PVBs) are frequently used for regional anesthesia for breast surgery. Ultrasound-guided paravertebral block is an advanced skill. The needle tip can be difficult to visualize with ultrasound, and the proximity to neurovascular structures as well as the pleura presents a risk of neurovascular injection and pneumothorax respectively. The midpoint transverse-process to pleura (MTP) block incorporates a novel needle endpoint that is technically easier to achieve and more distant from neurovascular structures and the pleura compared to traditional PVB. This study will compare the analgesic effects of MTP block to control and PVB.

ELIGIBILITY:
Inclusion Criteria:

* English or French Speaking
* Scheduled for major breast surgery
* ASA physical status classification I-III
* BMI <30kg/m2

Exclusion Criteria:

* Prior ipsilateral breast surgery
* Pre-existing neurological deficit or peripheral neuropathy involving the ipsilateral chest
* Contraindications to regional anesthesia
* Patient refusal of regional technique
* Chronic pain disorder
* Chronic opioid use
* Inability to provide informed consent

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative analgesia during the first 24 hours. | 48 hours
  Measured by opioid (equivalents of morphine) consumption and pain scores on a numerical rating scale.

SECONDARY OUTCOMES:
Post-operative quality of recovery during the first 24 hours. | 48 hours
  Measured by the Quality of recovery (QoR-15 scale).

CONTACTS AND LOCATIONS:
Overall Officials: Ioana Costache, MD, Principal Investigator — Ottawa Hospital, Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada